CLINICAL TRIAL: NCT07055490
Title: Effects of an Interdisciplinary Practice Bundle for Second-Stage of Labor on Clinical Outcomes
Brief Title: Interdisciplinary Practice Bundle for Second-Stage of Labor and Clinical Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Ahmed Fadel, Assis. professor of Woman's Health & Midwifery Nursing, Principal Investigator., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB. 0591
Record Dates: First submitted 2025-03-17; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Delivery Outcomes
Keywords: Bundle; Clinical outcomes; Second satge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apply interdisciplinary practice bundle during second-stage of labor (Experimental): interdisciplinary practices were combined in a bundle framework called (5-Ps) to maintain normal process during labor and prevent unnecessary routine interventions, which are (patience, positioning, physiological resuscitation, progress, and preventing urinary harm). These practices implemented from the beginning of the second stage of labor which is started from onset of complete cervical dilatation (10 cm) until delivery with a duration of 2 hours period.
  Interventions: Procedure: Interdisciplinary Practice Bundle
- control group (No Intervention): receive the routine hospital care

INTERVENTIONS:
Procedure: Interdisciplinary Practice Bundle — interdisciplinary practices were combined in a bundle framework called (5-Ps) to maintain normal process during labor and prevent unnecessary routine interventions, which are (patience, positioning, physiological resuscitation, progress, and preventing urinary harm). These practices implemented from the beginning of the second stage of labor which is started from onset of complete cervical dilatation (10 cm) until delivery with a duration of 2 hours period.
  Arms: Apply interdisciplinary practice bundle during second-stage of labor

SUMMARY:
This study aims to assess the effect of implementing an interdisciplinary practice bundle during second-stage of labor on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women aged greater than 18 years, with normal pregnancy.
* ≥ 38 weeks of gestation.
* Eligible for normal vaginal delivery

Exclusion Criteria:

* women with high risk pregnancy.
* Women with medical or psychological disorders.
* Women suspected to cesarean birth.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
1- Fatigue Visual Analogue Scale (VAS-F), | Study recruitment will take 6 months (from the beggining of July to the end of October, 2025) , all women who admitted to the labor and delivery unit at Mansoura University Hospitals, Egypt, were subjected to eligibility screening.
  Measurements I. Fatigue Visual Analogue Scale (VAS-F): a five point likert scale to assess fatigue post delivery.It is a self-reported scale consisted of 18 items relating to the subjective experience of fatigue with two subscales, fatigue (items 1-5 and 11-18) and energy (items 6-10). responces from "not at all tired" to "extremely tired". The total score calculated from sum of all items and categorized mild fatigue ranging from 0-3, moderate fatigue ranging from 4-6, and severe fatigue ranging from 7-10.
2- Childbirth Experience Questionnaire (CEQ) | Study recruitment will take 6 months (from the beggining of July to the end of October, 2025) , all women who admitted to the labor and delivery unit at Mansoura University Hospitals, Egypt, were subjected to eligibility screening.
  II. Childbirth Experience Questionnaire (CEQ). It is 22 items questionnaire yielded four domains (own capacity, perceived safety, professional support and participation.
  Scoring: Responses to 19 items were scored using a 4-point Likert scale ranging from 1 (totally disagree) to 4 (totally agree).